CLINICAL TRIAL: NCT00692341
Title: A Phase 1 Study To Evaluate The Pharmacokinetics Of AG-013736 In Subjects With Impaired Hepatic Function
Brief Title: Evaluation Of Hepatic Impairment On AG-013736 Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4061036
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Results first posted 2012-03-27 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Hepatic Insufficiency
Keywords: hepatic impairment
MeSH Terms: conditions — Hepatic Insufficiency | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hepatic Function - Mild Impairment (Experimental): Subjects with mild hepatic impairment (Child Pugh class A, score 5-6)
  Interventions: Drug: AG-013736
- Hepatic Function - Moderate Impairment (Experimental): Subjects with moderate hepatic impairment(Child Pugh class B,score 7-9)
  Interventions: Drug: AG-013736
- Hepatic Function - Normal (Experimental): Group 1
  1) subjects with normal hepatic function
  Interventions: Drug: AG-013736

INTERVENTIONS:
Drug: AG-013736 — Single oral 5-mg dose of AG-013736, administered as a film-coated, immediate-release tablet.
  Arms: Hepatic Function - Mild Impairment
Drug: AG-013736 — Single oral 5-mg dose of AG-013736, administered as a film-coated, immediate-release tablet.
  Arms: Hepatic Function - Moderate Impairment
Drug: AG-013736 — Single oral 5-mg dose of AG-013736, administered as a film-coated, immediate-release tablet.
  Arms: Hepatic Function - Normal

SUMMARY:
This study will evaluate the effects of mild and moderate impairment of hepatic function on the single-dose pharmacokinetics, safety and tolerability of AG-013736.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of reduced hepatic function (Child Pugh Classification A or B)
* Body Mass Index of 18-32 kg/m2

Exclusion Criteria:

* History of febrile illness within 5 days prior to first dose
* Any condition possibly affecting drug absorption (e.g. gastrectomy)
* Positive urine drug screen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Orlando, Florida

RESULTS

PARTICIPANT FLOW:
Groups:
- Axitinib : Normal Hepatic Function: Single oral dose of axitinib (AG-013736) 5 milligrams (mg) immediate release tablets (IRT) on Day 1 to participants with normal hepatic function.
- Axitinib : Mild Hepatic Impairment: Single oral dose of axitinib (AG-013736) 5 mg IRT on Day 1 to participants with mild hepatic impairment. Mild hepatic impairment (grade A) is defined as a Child-Pugh (CP) total score of 5-6. The CP classification assesses 5 hepatic parameters (total serum bilirubin, serum albumin, prothrombin time or prothrombin time international normalized ratio [INR], ascites and encephalopathy grade) on a scale of 1 (mild or none) to 3 (most severe). Total mild hepatic impairment score range is 5 (mild) to 15 (severe).
- Axitinib : Moderate Hepatic Impairment: Single oral dose of axitinib (AG-013736) 5 mg IRT on Day 1 to participants with moderate hepatic impairment. Moderate hepatic impairment (grade B) is defined as a CP total score of 7-9. The CP classification assesses 5 hepatic parameters (total serum bilirubin, serum albumin, prothrombin time or prothrombin time INR, ascites and encephalopathy grade) on a scale of 1 (mild or none) to 3 (most severe). Total moderate hepatic impairment score range is 5 (mild) to 15 (severe).
Period: Overall Study
Arm/Group | Axitinib : Normal Hepatic Function | Axitinib : Mild Hepatic Impairment | Axitinib : Moderate Hepatic Impairment
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Axitinib : Normal Hepatic Function | Axitinib : Mild Hepatic Impairment | Axitinib : Moderate Hepatic Impairment | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 47.4 (5.2) | 52.5 (5.6) | 54.3 (4.7) | 51.4 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 4
  Male | 7 | 7 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 12, 16, 24, 36, 48, 96 and 144 hours (hrs) post-dose
Population: Pharmacokinetic (PK) concentration population included all participants who were treated and had at least 1 concentration measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Axitinib : Normal Hepatic Function | Axitinib : Mild Hepatic Impairment | Axitinib : Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 8 | 8
ng/mL | 30.43 (50.00) | 26.96 (127.00) | 38.85 (50.00)
Statistical Analysis 1: Comparison: Axitinib : Normal Hepatic Function vs Axitinib : Mild Hepatic Impairment; For mild hepatic impairment, analysis of variance (ANOVA) was used to compare natural log transformed Cmax of axitinib (AG-013736) between the control group (normal hepatic function) and mild hepatic impairment. The point estimates and confidence intervals (CIs) on the log-scale were back transformed to provide estimates of the ratio of adjusted geometric means (mild hepatic impairment/normal hepatic function) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of adjusted geometric means = 88.61, 90% CI 2-sided [49.20 to 159.56]
Statistical Analysis 2: Comparison: Axitinib : Normal Hepatic Function vs Axitinib : Moderate Hepatic Impairment; For moderate hepatic impairment, ANOVA was used to compare natural log transformed Cmax of axitinib (AG-013736) between the control group (normal hepatic function) and moderate hepatic impairment. The point estimates and CIs on the log-scale were back transformed to provide estimates of the ratio of adjusted geometric means (moderate hepatic impairment/normal hepatic function) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of adjusted geometric means = 127.67, 90% CI 2-sided [70.90 to 229.91]

2. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)]
Description: AUC (0 - ∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 12, 16, 24, 36, 48, 96 and 144 hrs post-dose
Population: PK parameter analysis population included all participants who were treated and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Axitinib : Normal Hepatic Function | Axitinib : Mild Hepatic Impairment | Axitinib : Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 8 | 8
ng*hr/mL | 155.68 (63.00) | 121.96 (167.00) | 303.96 (44.00)
Statistical Analysis 1: Comparison: Axitinib : Normal Hepatic Function vs Axitinib : Mild Hepatic Impairment; For mild hepatic impairment, ANOVA was used to compare natural log transformed AUC (0 - ∞) of axitinib (AG-013736) between the control group (normal hepatic function) and mild hepatic impairment. The point estimates and CIs on the log-scale were back transformed to provide estimates of the ratio of adjusted geometric means (mild hepatic impairment/normal hepatic function) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of adjusted geometric means = 78.34, 90% CI 2-sided [39.92 to 153.75]
Statistical Analysis 2: Comparison: Axitinib : Normal Hepatic Function vs Axitinib : Moderate Hepatic Impairment; For moderate hepatic impairment, ANOVA was used to compare natural log transformed AUC (0 - ∞) of axitinib (AG-013736) between the control group (normal hepatic function) and moderate hepatic impairment. The point estimates and CIs on the log-scale were back transformed to provide estimates of the ratio of adjusted geometric means (moderate hepatic impairment/normal hepatic function) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of adjusted geometric means = 195.25, 90% CI 2-sided [99.49 to 383.18]

3. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast).
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 12, 16, 24, 36, 48, 96 and 144 hrs post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Axitinib : Normal Hepatic Function | Axitinib : Mild Hepatic Impairment | Axitinib : Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 8 | 8
ng*hr/mL | 148.43 (69.00) | 115.98 (180.00) | 295.23 (44.00)
Statistical Analysis 1: Comparison: Axitinib : Normal Hepatic Function vs Axitinib : Mild Hepatic Impairment; For mild hepatic impairment, ANOVA was used to compare natural log transformed AUClast of axitinib (AG-013736) between the control group (normal hepatic function) and mild hepatic impairment. The point estimates and CIs on the log-scale were back transformed to provide estimates of the ratio of adjusted geometric means (mild hepatic impairment/normal hepatic function) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of adjusted geometric means = 78.14, 90% CI 2-sided [38.68 to 157.82]
Statistical Analysis 2: Comparison: Axitinib : Normal Hepatic Function vs Axitinib : Moderate Hepatic Impairment; For moderate hepatic impairment, ANOVA was used to compare natural log transformed AUClast of axitinib (AG-013736) between the control group (normal hepatic function) and moderate hepatic impairment. The point estimates and CIs on the log-scale were back transformed to provide estimates of the ratio of adjusted geometric means (moderate hepatic impairment/normal hepatic function) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of adjusted geometric means = 198.90, 90% CI 2-sided [98.47 to 401.74]

4. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 12, 16, 24, 36, 48, 96 and 144 hrs post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | Axitinib : Normal Hepatic Function | Axitinib : Mild Hepatic Impairment | Axitinib : Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 8 | 8
hr | 3.50 [2.00 to 4.00] | 2.75 [1.00 to 4.00] | 4.00 [1.50 to 4.00]

5. Secondary Outcome: Plasma Elimination Half-life (t1/2)
Description: Plasma elimination half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 12, 16, 24, 36, 48, 96 and 144 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Axitinib : Normal Hepatic Function | Axitinib : Mild Hepatic Impairment | Axitinib : Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 8 | 8
hr | 4.74 (3.77) | 3.61 (3.02) | 7.12 (6.49)

6. Secondary Outcome: Apparent Oral Clearance (CL/F)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the oral bioavailability. Clearance was estimated from population PK modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 12, 16, 24, 36, 48, 96 and 144 hrs post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Axitinib : Normal Hepatic Function | Axitinib : Mild Hepatic Impairment | Axitinib : Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 8 | 8
mL/min | 535.3 (63.0) | 683.3 (167.0) | 274.2 (44.0)

7. Secondary Outcome: Apparent Volume of Distribution (Vz/F)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the oral bioavailability.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 12, 16, 24, 36, 48, 96 and 144 hrs post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Axitinib : Normal Hepatic Function | Axitinib : Mild Hepatic Impairment | Axitinib : Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 8 | 8
Liter (L) | 166.43 (52.00) | 162.65 (87.00) | 127.68 (67.00)

8. Secondary Outcome: Fraction of Unbound Drug (fu)
Description: Fraction of unbound drug (fu) is defined as the ratio of unbound drug concentration to the total drug concentration.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 12, 16, 24, 36, 48, 96 and 144 hrs post-dose
Population: PK parameter analysis population included all participants who were treated and had at least 1 of the PK parameters of interest. Here, the 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure for each group respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Axitinib : Normal Hepatic Function | Axitinib : Mild Hepatic Impairment | Axitinib : Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 5 | 8
Ratio | 0.004 (25.000) | 0.003 (50.000) | 0.004 (134.000)
Statistical Analysis 1: Comparison: Axitinib : Normal Hepatic Function vs Axitinib : Mild Hepatic Impairment; For mild hepatic impairment, ANOVA was used to compare natural log transformed fu of axitinib (AG-013736) between the control group (normal hepatic function) and mild hepatic impairment. The point estimates and CIs on the log-scale were back transformed to provide estimates of the ratio of adjusted geometric means (mild hepatic impairment/normal hepatic function) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of adjusted geometric means = 73.78, 90% CI 2-sided [37.40 to 145.56]
Statistical Analysis 2: Comparison: Axitinib : Normal Hepatic Function vs Axitinib : Moderate Hepatic Impairment; For moderate hepatic impairment, ANOVA was used to compare natural log transformed fu of axitinib (AG-013736) between the control group (normal hepatic function) and moderate hepatic impairment. The point estimates and CIs on the log-scale were back transformed to provide estimates of the ratio of adjusted geometric means (moderate hepatic impairment/normal hepatic function) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of adjusted geometric means = 100.86, 90% CI 2-sided [55.58 to 183.02]

9. Secondary Outcome: Unbound Apparent Oral Clearance (CLu/F)
Description: Clearance of an unbound drug is a measure of the rate at which an unbound drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the oral bioavailability. Unbound drug clearance is a quantitative measure of the rate at which an unbound drug substance is removed from the blood.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 12, 16, 24, 36, 48, 96 and 144 hrs post-dose
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Axitinib : Normal Hepatic Function | Axitinib : Mild Hepatic Impairment | Axitinib : Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 5 | 8
mL/min | 132218.6 (56.0) [10000 to 16000] | 120883.5 (82.0) [9000 to NA] | 67143.1 (109.0)
Statistical Analysis 1: Comparison: Axitinib : Normal Hepatic Function vs Axitinib : Mild Hepatic Impairment; For mild hepatic impairment, ANOVA was used to compare natural log transformed CLu/F of axitinib (AG-013736) between the control group (normal hepatic function) and mild hepatic impairment. The point estimates and CIs on the log-scale were back transformed to provide estimates of the ratio of adjusted geometric means (mild hepatic impairment/normal hepatic function) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of adjusted geometric means = 91.43, 90% CI 2-sided [44.75 to 186.79]
Statistical Analysis 2: Comparison: Axitinib : Normal Hepatic Function vs Axitinib : Moderate Hepatic Impairment; For moderate hepatic impairment, ANOVA was used to compare natural log transformed CLu/F of axitinib (AG-013736) between the control group (normal hepatic function) and moderate hepatic impairment. The point estimates and CIs on the log-scale were back transformed to provide estimates of the ratio of adjusted geometric means (moderate hepatic impairment/normal hepatic function) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of adjusted geometric means = 50.78, 90% CI 2-sided [27.14 to 95.03]

10. Secondary Outcome: Unbound Apparent Volume of Distribution (Vzu/F)
Description: Volume of distribution of unbound drug is defined as the theoretical volume in which the total amount of unbound drug would need to be uniformly distributed to produce the desired plasma concentration of unbound drug. Unbound apparent volume of distribution after oral dose (Vzu/F) is influenced by the oral bioavailability.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 12, 16, 24, 36, 48, 96 and 144 hrs post-dose
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Axitinib : Normal Hepatic Function | Axitinib : Mild Hepatic Impairment | Axitinib : Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 5 | 8
L | 41108.6 (57.0) | 42378.3 (40.0) | 31268.8 (121.0)
Statistical Analysis 1: Comparison: Axitinib : Normal Hepatic Function vs Axitinib : Mild Hepatic Impairment; For mild hepatic impairment, ANOVA was used to compare natural log transformed Vzu/F of axitinib (AG-013736) between the control group (normal hepatic function) and mild hepatic impairment. The point estimates and CIs on the log-scale were back transformed to provide estimates of the ratio of adjusted geometric means (mild hepatic impairment/normal hepatic function) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of adjusted geometric means = 103.09, 90% CI 2-sided [51.53 to 206.22]
Statistical Analysis 2: Comparison: Axitinib : Normal Hepatic Function vs Axitinib : Moderate Hepatic Impairment; For moderate hepatic impairment, ANOVA was used to compare natural log transformed Vzu/F of axitinib (AG-013736) between the control group (normal hepatic function) and moderate hepatic impairment. The point estimates and CIs on the log-scale were back transformed to provide estimates of the ratio of adjusted geometric means (moderate hepatic impairment/normal hepatic function) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of adjusted geometric means = 76.06, 90% CI 2-sided [41.41 to 139.73]

11. Secondary Outcome: Unbound Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)u]
Description: AUC (0 - ∞)u = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞) for unbound drug. It is obtained from AUCu (0 - t) plus AUCu (t - ∞).
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 12, 16, 24, 36, 48, 96 and 144 hrs post-dose
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Axitinib : Normal Hepatic Function | Axitinib : Mild Hepatic Impairment | Axitinib : Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 5 | 8
ng*hr/mL | 0.63 (56.00) | 0.69 (82.00) | 1.24 (109.00)
Statistical Analysis 1: Comparison: Axitinib : Normal Hepatic Function vs Axitinib : Mild Hepatic Impairment; For mild hepatic impairment, ANOVA was used to compare natural log transformed AUC (0 - ∞)u of axitinib (AG-013736) between the control group (normal hepatic function) and mild hepatic impairment. The point estimates and CIs on the log-scale were back transformed to provide estimates of the ratio of adjusted geometric means (mild hepatic impairment/normal hepatic function) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of adjusted geometric means = 109.38, 90% CI 2-sided [53.54 to 223.47]
Statistical Analysis 2: Comparison: Axitinib : Normal Hepatic Function vs Axitinib : Moderate Hepatic Impairment; For moderate hepatic impairment, ANOVA was used to compare natural log transformed AUC (0 - ∞)u of axitinib (AG-013736) between the control group (normal hepatic function) and moderate hepatic impairment. The point estimates and CIs on the log-scale were back transformed to provide estimates of the ratio of adjusted geometric means (moderate hepatic impairment/normal hepatic function) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of adjusted geometric means = 196.92, 90% CI 2-sided [105.23 to 368.49]

12. Secondary Outcome: Unbound Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClastu)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClastu) for unbound drug.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 12, 16, 24, 36, 48, 96 and 144 hrs post-dose
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Axitinib : Normal Hepatic Function | Axitinib : Mild Hepatic Impairment | Axitinib : Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 5 | 8
ng*hr/mL | 0.60 (61.00) | 0.67 (81.00) | 1.21 (106.00)
Statistical Analysis 1: Comparison: Axitinib : Normal Hepatic Function vs Axitinib : Mild Hepatic Impairment; For mild hepatic impairment, ANOVA was used to compare natural log transformed AUClastu of axitinib (AG-013736) between the control group (normal hepatic function) and mild hepatic impairment. The point estimates and CIs on the log-scale were back transformed to provide estimates of the ratio of adjusted geometric means (mild hepatic impairment/normal hepatic function) and 90% CIs for the ratios; Test type: Superiority or Other; Adjusted ratio of geometric means = 111.65, 90% CI 2-sided [54.35 to 229.37]
Statistical Analysis 2: Comparison: Axitinib : Normal Hepatic Function vs Axitinib : Moderate Hepatic Impairment; For moderate hepatic impairment, ANOVA was used to compare natural log transformed AUClastu of axitinib (AG-013736) between the control group (normal hepatic function) and moderate hepatic impairment. The point estimates and CIs on the log-scale were back transformed to provide estimates of the ratio of adjusted geometric means (moderate hepatic impairment/normal hepatic function) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of adjusted geometric means = 200.60, 90% CI 2-sided [106.68 to 377.20]

13. Secondary Outcome: Unbound Maximum Observed Plasma Concentration (Cmaxu)
Description: Cmaxu is the highest measured unbound plasma concentration during the dosing interval.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 12, 16, 24, 36, 48, 96 and 144 hrs post-dose
Population: PK concentration population included all participants who were treated and had at least 1 concentration measurement. Here, the 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure for each group respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Axitinib : Normal Hepatic Function | Axitinib : Mild Hepatic Impairment | Axitinib : Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 5 | 8
ng/mL | 0.12 (46.00) | 0.13 (47.00) | 0.16 (97.00)
Statistical Analysis 1: Comparison: Axitinib : Normal Hepatic Function vs Axitinib : Mild Hepatic Impairment; For mild hepatic impairment, ANOVA was used to compare natural log transformed Cmaxu of axitinib (AG-013736) between the control group (normal hepatic function) and mild hepatic impairment. The point estimates and CIs on the log-scale were back transformed to provide estimates of the ratio of adjusted geometric means (mild hepatic impairment/normal hepatic function) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of adjusted geometric means = 106.82, 90% CI 2-sided [58.22 to 195.99]
Statistical Analysis 2: Comparison: Axitinib : Normal Hepatic Function vs Axitinib : Moderate Hepatic Impairment; For moderate hepatic impairment, ANOVA was used to compare natural log transformed Cmaxu of axitinib (AG-013736) between the control group (normal hepatic function) and moderate hepatic impairment. The point estimates and CIs on the log-scale were back transformed to provide estimates of the ratio of adjusted geometric means (moderate hepatic impairment/normal hepatic function) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of adjusted geometric means = 128.76, 90% CI 2-sided [75.62 to 219.25]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Axitinib : Normal Hepatic Function | Axitinib : Mild Hepatic Impairment | Axitinib : Moderate Hepatic Impairment
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/8 | 0/8 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib : Normal Hepatic Function (N=8) | Axitinib : Mild Hepatic Impairment (N=8) | Axitinib : Moderate Hepatic Impairment (N=8)
Headache (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.